CLINICAL TRIAL: NCT00971516
Title: Healing Profile of Titanium Dental Implants Placed in Patients With Type 2 Diabetes: a Prospective Osteoimmunological and Clinical Pilot Study
Brief Title: Healing Profile of Titanium Dental Implants Placed in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Collaborators: University of Manitoba (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Getulio Nogueira, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPL900209-01
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes; Dental Implants
Keywords: diabetes; implants; cytokines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes (Active Comparator): compare cytokines between diabetes and non diabetes patients
  Interventions: Procedure: Implants surgery
- Implants (Active Comparator): Compare implant healing phases
  Interventions: Procedure: Implant placement; Procedure: Implants surgery

INTERVENTIONS:
Procedure: Implant placement — dental implant placement
  Other Names: Dental implants
  Arms: Implants
Procedure: Implants surgery — dental implant surgery
  Other Names: diabetes patients

SUMMARY:
The main goal of this study is to look at the way gums heal around dental implants placed in healthy patients compared to patients with type 2 diabetes. This study is designed to answer the following questions:

* How much swelling occurs around dental implants placed in patients with type 2 diabetes?
* Is swelling (inflammation) present or absent in the initial healing phase after placement of dental implants?
* What are the differences in the amount of swelling (inflammation) in patients with and without type 2 diabetes? Are patients with type 2 diabetes more likely to have bone loss around dental implants?

DETAILED DESCRIPTION:
Rationale:

For the evaluation/ monitoring of dental implants, practitioners seem to use simultaneously a variety of the clinical, image-based and laboratory measurements, probably because of the fact that each of these measures is likely to provide important information regarding the complex series of events at the dental implant sites (Guncu et al 2008). Thus, the proposed study seeks to characterize for the first time, the healing profile of dental implants in type 2 diabetic patients when compared with natural teeth, in the lights of the microarray quantitative evaluation of the host response promoted by cytokines and osteoclastogenesis-related factors levels, and correlates the quantitative findings with qualitative high-tech multi-modal clinical infra-red diagnosis data. This information may allow the development of new therapeutic intervention modalities to maximize the protective and minimize the destructive aspects of inflammation in peri-implant tissues even in early stages. If the results of this preliminary study are positive, a longitudinal follow-up study will be conducted within the same population to investigate this relationship over a long-term period.

Methods:

A 1-year prospective pilot study will be performed in 20 patients (males; 35-55 year old), 10 controlled type 2 diabetics (HbA1c values < 7.2%) and 10 non diabetics matched for implant treatment indications to serve as controls (all suffering from partial edentulism). Patients will receive at least one dental implant (Ankylos®, Dentsply, Germany). Patients attending the Graduate Periodontics Clinic (University of Manitoba) will be invited to participate in the study. A comprehensive history will be taken and an examination of the oral cavity will be carried out for each patient for implant evaluation. Based on a review of the history and the examination findings by one of the study personnel, potential subjects will be identified who satisfy the following inclusion and exclusion criteria. Excluded from the study will be those with active periodontal disease, uncontrolled diabetes, smokers, any metabolic bone diseases or other systemic disorders. All patients will be informed about the nature of the study and volunteers will sign an informed consent form prior to entry into the study. The patients will receive at least 1 one-stage Ankylos® implant (Dentsply, Germany) in the same bone area. After restoration, the patients will be followed up for up to 1 year. The healing profile will be determined quantitatively by cytokines and biomarkers in peri-implant crevicular fluid (PICF) (microarray) and qualitatively by the inflammatory infiltrate (IR evaluation).

Aims and Approaches:

Aim 1- To establish quantitatively and qualitatively the healing profile of dental implants placed in type 2 diabetic patients.

Aim 2- To compare the levels of cytokines between dental implants and natural teeth.

Approach: PICF/GCF samples will be collected from diabetic and non diabetic patients. The volume of PICF/GCF will be determined (Periotron 8000®) for subsequent cytokine assays (Schierano et al 2008). All samples will be evaluated simultaneously by microarray technique (Genepix®) for quantitative measurement of the concentration of multiple cytokines: IL-1β, IL-2, IL-4, IL-6, IL-8, TNF-α, IFN-γ, IL-10, IL-12p70, IL-13, TGF-β, IL-17 and IL-23, as well as OPG and RANK-L; qualitative measurements will be performed by infra-red diagnosis.

Aim 3- To determine the initial bone stability of dental implants placed in diabetic patients.

Approach: Statistical analysis will correlate all data from many time points regarding the cytokine levels from implants and teeth (PICF/GCF respectively) and from all patients (diabetics and non diabetics) to verify the impact of host response on inflammation and bone stability over time.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients and with partial edentulism.

Exclusion Criteria:

* Active periodontal disease,
* Uncontrolled diabetes,
* Smokers,
* Any metabolic bone diseases or other systemic disorders.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Healing profile of cytokines | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Getulio R Nogueira F, Principal Investigator — University of Manitoba